CLINICAL TRIAL: NCT03233269
Title: BEATS 2: The Effects of Music Therapy on Young Adults With Sickle Cell Disease
Brief Title: BEATS 2: Music Therapy in Sickle Cell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Kulas Foundation (Other)
Responsible Party: Principal Investigator, Samuel Rodgers-Melnick, Music Therapist-Board Certified, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-17-07
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music Therapy Group (Experimental): Music therapy is the clinical and evidence-based use of music interventions to accomplish individualized goals within a therapeutic relationship by a credentialed professional who has completed an approved music therapy program. Music therapy is an established health profession in which music is used within a therapeutic relationship to address physical, emotional, cognitive, and social needs of individuals (American Music Therapy Association [AMTA], 2013, para 1 and 2).
  Interventions: Behavioral: Music Therapy

INTERVENTIONS:
Behavioral: Music Therapy — During the educational music therapy intervention, member(s) of the Adult Sickle Cell Disease team will share with the patients the medical information pertinent to the appointment via a prerecorded video. The Music Therapist will then engage the patients in a music therapy intervention designed to teach and reinforce the skills and knowledge presented. These music therapy interventions may include but are not limited to original songs/rap/instrumental playing, vocal and/or instrumental improvisation, patient-contributed lyrics, mnemonics, and stress and pain reducing strategies. The music therapy interventions will be tailored to best convey the educational message.

SUMMARY:
The purpose of this study is to investigate the effects of the BEATS music therapy program on the self-efficacy, trust, knowledge, and adherence of young adult patients with SCD.

Primary Hypotheses:

Compared to baseline, young adult patients with SCD who receive the music therapy interventions will report:

Higher sickle cell self-efficacy as measured by the Sickle Cell Self Efficacy Scale (SCSES), Higher trust in health care providers as measured by the Wake Forest Trust in the Medical Profession Scale, and Higher SCD knowledge as measured by the Seidman Sickle Cell Knowledge Quiz.

Secondary Hypotheses Compared to the one year prior to the study period, young adults with SCD who receive the music therapy interventions will have a higher rate of adherence to clinic appointments during the one-year study period.

Additional Questions Do music therapy interventions influence the rate of hospital utilization as measured by ED visits, Acute Care Clinic (ACC) visits, and admissions during the study period compared to the previous year? Do music therapy interventions influence adherence to hydroxyurea therapy for patients receiving hydroxyurea as measured by change in mean corpuscular volume (MCV) during the study period? Do music therapy interventions influence adherence to iron chelation therapy for patients receiving iron chelation therapy as measured by ferritin count during the study period? Does the schedule of music therapy interventions in this study improve outcomes more significantly than the schedule of music therapy interventions from [IRB# 03-15-30]?

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 35 years of age
* Subject is diagnosed with sickle cell disease
* Subject is able to speak and understand English
* Subject has a working email address.
* Subject has access to a mobile device with email capabilities.

Exclusion Criteria:

* Subject has significant hearing impairment that has not been corrected
* Subject has significant visual impairment that has not been corrected

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in scores on the Sickle Cell Self-Efficacy Scale (SCSES) | Baseline, immediately after session 4, 4 weeks after session 4, immediately after session 8, 4 weeks after session 8.
  Self-efficacy is the conviction that one can successfully execute the behavior required to produce the outcome.
  (Bandura, 1997, p. 193). The SCSES is a nine-item Likert scale originally developed for adults with sickle cell disease (Edwards, Telfair, Cecil, & Lenoci, 2000) and revised in a follow up study by Clay and Telfair (2007) for adolescents using a sample of 131 individuals age 11-19.
Change from baseline in scores on the Wake Forest Trust in the Medical Profession Scale | Baseline, immediately after session 4, 4 weeks after session 4, immediately after session 8, 4 weeks after session 8.
  Patient trust is the optimistic acceptance of a vulnerable situation in which the patient believes the health-care provider will take care of the patient's interests (Dugan, Trachtenberg, & Hall, 2005).The Wake Forest Trust in the Medical Profession Scale is a five-item scale in which respondents express their level of agreement with the following statements: 1) Sometimes doctors care more about what is convenient for them than about their patients' medical needs (reverse coded); 2) Doctors are extremely thorough and careful; 3) You completely trust doctors' decisions about which medical treatments are best; 4) A doctor would never mislead you about anything; 5) All in all, you trust your doctor completely. Responses are summed and scores are on a 5-25 scale, with higher values indicating greater trust.
Change from baseline in scores on the Seidman Sickle Cell Knowledge Quiz | Baseline, immediately after session 4, 4 weeks after session 4, immediately after session 8, 4 weeks after session 8.
  Sickle Cell Disease knowledge will be measured using the Seidman Sickle Cell Knowledge Quiz developed specifically for this study. The Seidman Sickle Cell Knowledge Quiz is adapted from questions from the Sickle Cell Disease Knowledge Test (Kaslow et al., 2000) and How Much Do I Know About Sickle Cell Disease (Baskin, Collins, Kaslow, & Hsu, 2002).

SECONDARY OUTCOMES:
Change from baseline in rate of adherence to clinic appointments during the one-year study period. | Baseline, 12 months
  Adherence is the extent to which a person's behavior coincides with medical or prescribed health advice (Julius, 2009).Adherence will be measured regularly throughout the study via medical record review. In order to assess adherence, the following data will be obtained from the medical record on each patient throughout the study period: 1) Total scheduled clinic visits with Adult Sickle Cell Disease Clinic, 2) Number of missed clinic visits to Adult Sickle Cell Disease Clinic due to no show, cancellation, or rescheduling

CONTACTS AND LOCATIONS:
Overall Officials: Samuel N Rodgers-Melnick, MT-BC, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals Seidman Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- See also: Website for music therapy program at UH Seidman Cancer Center — http://www.uhseidman.org/musictherapy